CLINICAL TRIAL: NCT02986672
Title: ADHD and Nutrition: The Influence of Omega-3 on ADHD Related Symptoms
Brief Title: Intervention With Omega-3 in Children With Attention Deficit Hyperactivity Disorder(ADHD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADHD_Kvernmo
Record Dates: First submitted 2016-01-08; First posted 2016-12-08 (Estimated); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: ADHD; ADD
Keywords: ADHD; omega 3; children; nutrition; MUFA; ADD; PUFA; Calanus; learning difficulties
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Calanus oil (Active Comparator): Children receiving omega-3 in form om calanus oil in capsule form
  Interventions: Dietary Supplement: Calanus oil
- Placebo (Placebo Comparator): Children receiving medical paraffin in capsule form (2 ml volume per day)
  Interventions: Other: Medical Paraffin

INTERVENTIONS:
Dietary Supplement: Calanus oil — Omega-3 oil in form of calanus oil
  Arms: Calanus oil
Other: Medical Paraffin — 2ml per day
  Arms: Placebo

SUMMARY:
This study aims to determine if marine monounsaturated and polyunsaturated fatty acids can benefit children aged 6-16 years with ADHD and related symptoms. It is a randomized, double-blind, placebo-controlled study involving approximately 330 children from Norway. The study will assess ADHD symptoms reported by caregivers, teachers, and the child at baseline, after 6 months of treatment, and 6 months post-treatment. Secondary outcomes will include reading and writing difficulties, cognitive functions, and physical health.

DETAILED DESCRIPTION:
Children with ADHD often exhibit low blood levels of omega-3 fatty acids, which are not correlated with their diet. Low omega-3 levels are associated with poor cognition and behavior. Previous research indicates that omega-3 supplements can enhance literacy, behavior, memory, and reaction time in children with ADHD, although the improvements are generally small to modest.

A study on adolescent mental health in North Norway from 2003-2005 revealed that adolescents consuming more fish had lower levels of hyperactivity compared to those with lower fish consumption (unpublished results from The Norwegian Arctic Adolescent Health Study, Siv Kvernmo).

Key limitations in existing studies include small sample sizes, varying methodologies, short intervention periods, and the absence of control groups. This study addresses these limitations by using whole marine oil from the zooplankton Calanus finmarchicus, which naturally contains stearidonic acid (a precursor to EPA) and astaxanthin, a natural antioxidant.

Previous clinical studies did not utilize pure oil from zooplankton such as Calanus finmarchicus. This oil is not chemically processed, retaining its natural antioxidants.

Blood tests will be conducted before and after the 6-month intervention period to measure the omega-3 index and include general hematology and biochemistry.

ELIGIBILITY:
Inclusion Criteria:

- ADHD according to DSM-IV criteria

Exclusion Criteria:

* IQ below 70
* infantil autism, psychosis, bipolar disorders and serious somatic disease
* any abnormal or pathological blood test during trial
* ADHD medication

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 332 (Actual)
Dates: Start 2017-11-03 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-09-20 (Actual)

PRIMARY OUTCOMES:
Swanson, Nolan, and Pelham IV Questionnaire | 0, 3, 6, and 12 months
  Description: The SNAP-IV is a 90-item scale used to evaluate symptoms of ADHD and related disorders.
  Score Range: Minimum value: 0, Maximum value: 270 Interpretation: Higher scores indicate worse symptoms.

SECONDARY OUTCOMES:
Behavior Rating Inventory of Executive Function | 0, 3, 6, and 12 months
  Description: The BRIEF assesses executive function behaviors in children and adolescents in home and school environments.
  Score Range: Minimum value: 0, Maximum value: 240 Interpretation: Higher scores indicate worse executive function behaviors.
ADHD Rating Scale by Russell Barkley | 0, 3, 6, and 12 months
  Reduction in symptom score. Reduction in symptom score. Minimum value: 0, Maximum value: 54. Higher scores
Affective Reactivity Index | 0, 3, 6, and 12 months
  Description: The ARI is a scale that measures irritability, consisting of six symptom items and one impairment item.
  Score Range: Minimum value: 0, Maximum value: 12 Interpretation: Higher scores indicate greater irritability.
Test of Variables of Attention | 0, 3, 6, and 12 months
  Description: The TOVA is a computerized test that measures attention-related problems in individuals aged 8 years and older.
  Score Range: Minimum value: -10, Maximum value: 10 Interpretation: Higher scores indicate better attention performance.
Strengths and Difficulties Questionnaire | 0, 3, 6, and 12 months
  Description: The SDQ is a psychological screening tool used to assess the behavioral and emotional strengths and difficulties of children and adolescents, consisting of 25 items across five dimensions.
  Score Range: Minimum value: 0, Maximum value: 50 Interpretation: Higher scores indicate more behavioral and emotional difficulties.
KIDSCREEN-52 | 0, 3, 6, and 12 months
  Description: The KIDSCREEN-52 is a questionnaire that examines Health-Related Quality of Life (HRQoL) in children and adolescents, consisting of 52 items.
  Score Range: Minimum value: 52, Maximum value: 260 Interpretation: Higher scores indicate better health-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Siv Kvernmo, MD PhD, Study Director — University of Tromso
Locations (2):
- Norway (2):
  - Finnmarkssykehuset SANKS BUP Karasjok, Karasjok, Finnmark Fylke
  - University Hospital of North Norway, Tromsø, Troms

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Raine A, Portnoy J, Liu J, Mahoomed T, Hibbeln JR. Reduction in behavior problems with omega-3 supplementation in children aged 8-16 years: a randomized, double-blind, placebo-controlled, stratified, parallel-group trial. J Child Psychol Psychiatry. 2015 May;56(5):509-20. doi: 10.1111/jcpp.12314. Epub 2014 Aug 22. PMID 25146492
- [Background] Gow RV, Hibbeln JR, Parletta N. Current evidence and future directions for research with omega-3 fatty acids and attention deficit hyperactivity disorder. Curr Opin Clin Nutr Metab Care. 2015 Mar;18(2):133-8. doi: 10.1097/MCO.0000000000000140. PMID 25581035
- [Background] Heilskov Rytter MJ, Andersen LB, Houmann T, Bilenberg N, Hvolby A, Molgaard C, Michaelsen KF, Lauritzen L. Diet in the treatment of ADHD in children - a systematic review of the literature. Nord J Psychiatry. 2015 Jan;69(1):1-18. doi: 10.3109/08039488.2014.921933. Epub 2014 Jun 16. PMID 24934907
- [Background] Milte CM, Sinn N, Buckley JD, Coates AM, Young RM, Howe PR. Polyunsaturated fatty acids, cognition and literacy in children with ADHD with and without learning difficulties. J Child Health Care. 2011 Dec;15(4):299-311. doi: 10.1177/1367493511403953. Epub 2011 Aug 9. PMID 21828168
- [Background] Stonehouse W, Conlon CA, Podd J, Hill SR, Minihane AM, Haskell C, Kennedy D. DHA supplementation improved both memory and reaction time in healthy young adults: a randomized controlled trial. Am J Clin Nutr. 2013 May;97(5):1134-43. doi: 10.3945/ajcn.112.053371. Epub 2013 Mar 20. PMID 23515006
- [Background] Richardson AJ. Omega-3 fatty acids in ADHD and related neurodevelopmental disorders. Int Rev Psychiatry. 2006 Apr;18(2):155-72. doi: 10.1080/09540260600583031. PMID 16777670
- [Background] Montgomery P, Burton JR, Sewell RP, Spreckelsen TF, Richardson AJ. Low blood long chain omega-3 fatty acids in UK children are associated with poor cognitive performance and behavior: a cross-sectional analysis from the DOLAB study. PLoS One. 2013 Jun 24;8(6):e66697. doi: 10.1371/journal.pone.0066697. Print 2013. PMID 23826114
- [Background] Hoper AC, Salma W, Sollie SJ, Hafstad AD, Lund J, Khalid AM, Raa J, Aasum E, Larsen TS. Wax esters from the marine copepod Calanus finmarchicus reduce diet-induced obesity and obesity-related metabolic disorders in mice. J Nutr. 2014 Feb;144(2):164-9. doi: 10.3945/jn.113.182501. Epub 2013 Nov 27. PMID 24285691
- [Background] Eilertsen KE, Maehre HK, Jensen IJ, Devold H, Olsen JO, Lie RK, Brox J, Berg V, Elvevoll EO, Osterud B. A wax ester and astaxanthin-rich extract from the marine copepod Calanus finmarchicus attenuates atherogenesis in female apolipoprotein E-deficient mice. J Nutr. 2012 Mar;142(3):508-12. doi: 10.3945/jn.111.145698. Epub 2012 Feb 8. PMID 22323762
- [Derived] Gillies D, Leach MJ, Perez Algorta G. Polyunsaturated fatty acids (PUFA) for attention deficit hyperactivity disorder (ADHD) in children and adolescents. Cochrane Database Syst Rev. 2023 Apr 14;4(4):CD007986. doi: 10.1002/14651858.CD007986.pub3. PMID 37058600